CLINICAL TRIAL: NCT05787717
Title: Parental Presence at Anesthesia Induction in Infants - a Randomized Controlled Trial
Brief Title: Parental Presence at Anesthesia Induction
Acronym: PPAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Peter Frykholm, Principal Investigator, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PPAI1
Record Dates: First submitted 2023-02-23; First posted 2023-03-28 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Parent-Child Relations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental presence (Experimental): Parents are present and active in the care of their child until general anesthesia has been established in the operating room
  Interventions: Other: Parental presence
- Control (No Intervention): Parents leave their infant in the holding area of the operating rooms

INTERVENTIONS:
Other: Parental presence — The parent is encouraged to stay close to their child and are given ample room on one side of the OR table for this purpose
  Arms: Parental presence

SUMMARY:
Parental presence during induction for young infants is still debated. There is a paucity of information on the real-world interaction between parents, infant and the anesthesia team.

Aim To investigate parents' anxiety, need of information and experiences during induction of their infant, as well as staff communication and experiences, using quantitative and qualitative methods.

Methods Randomized controlled trial of parent´s experiences of participating in their infant´s anesthesia induction. Parents will be randomized to being present in the operating room until the infant is asleep due to anesthesia induction (intervention group), or leaving their child to the anesthesia team in the OR holding area (control group).

DETAILED DESCRIPTION:
Background Surgery in a paediatric setting involves a considerable amount of stress for children and for their parents. The pros and cons of parental presence during anesthesia induction are debated, especially in infants. In older children, parents play a critical role in paediatric surgery, since children depend on parents for support and guidance in coping. However, many centers will not allow parental presence for young infants and neonates, since attachment relationships develop during the second half of infancy (6 - 12 months of age), and the risk of complications during induction are increased. However, there is a paucity of information on the real-world interaction between parents, infant and the anesthesia team. Therefore, the present study will investigate how parental presence affects the parents´ perioperative anxiety level and experiences in a randomized controlled trial. Anesthesia team communication, attitudes and experiences and the rate of complications during induction and emergence will also be studied. The study hypothesis is that presence at induction reduces the parents' anxiety level.

Aim To investigate parents' anxiety, need of information and experiences during induction of their infant, as well as staff communication and experiences, using quantitative and qualitative methods.

Methods Design: randomized controlled trial. After informed consent has been obtained from both parents, they are randomized to being present in the operating room until the infant is asleep due to anesthesia induction (intervention group), or leaving their child to the anesthesia team in the Operating Room (OR)holding area (control group).

When they arrive at the OR holding area, the parents are asked to fill in the Amsterdam Preoperative Anxiety and Information Scale (APAIS) questionnaire. Electrocardiogram (EKG) electrodes are placed on the infant's chest and connected to an anesthesia monitor. Then the infant is transported to the OR together with the parent if in the intervention group. In the intervention group, the parent is encouraged to stay close to their child and are given ample room on one side of the OR table for this purpose. If appropriate, a peripheral i.v. line is placed. A standard pre-induction time-out is performed, after which the anesthesia induction starts (i.v. thiopental or propofol if a line is in place, mask induction with sevoflurane if not). As soon as the child is asleep (no voluntary movements, eyes closed), the parents are escorted out of the OR, and are asked to fill in the APAIS questionnaire a second time. As in the control group, they are informed that they will be called to the Post Anesthesia Care Unit (PACU) at the end of the procedure.

Depending on investigator availability, the parents will be interviewed about their experiences on the day after surgery. In addition, the nurse anesthetist and attending anesthesiologist will be interviewed on the day of surgery.

The induction and the emergence will be video recorded and field notes will be taken by a separate investigator taking care not to disturb the procedure.

Field notes, video-recordings and interviews will be transcribed and analyzed using phenomenological/hermeneutic methods. Open questions about how the subject experienced the induction will be posed, and follow-up questions to obtain in-depth understanding of the subjects' sentiments and reflections.

ELIGIBILITY:
Inclusion Criteria:

* Infant scheduled for general anesthesia
* parents are available, accompanying their infant

Exclusion Criteria:

* age of infant > 6 months
* critical illness (supplementary oxygen, inotropic support or ventilator therapy)

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
APAIS Anxiety | Within 5 minutes of leaving their child to the anesthesia team.
  Parents fill out the form Amsterdam Preoperative Anxiety and Information Scale. The Anxiety component of the scale har four items and the total score (minimum value 4, max 20) is the primary outcome. High scores indicate worse outcome.

SECONDARY OUTCOMES:
Infant´s heart rate | From when EKG monitoring starts in the holding area until child is unresponsive due to general anesthesia - a time fram of up to 15 minutes
  The changes in heart rate of the infant during the pre-induction period and during induction.
Adverse events | Anesthesia induction (a time frame of up to 10 minutes)
  Adverse events during induction such as desaturation, bradycardia, hypotension, difficult intubation, difficult i.v. access.
Staff interview data | Within 24 hours after the case is finished in the OR
  The staff self-reported experience of parental presence at induction (interview data)
Parental interview data | Within 48 hours after the case is finished in the OR
  The parents self-reported experience of leaving their child before surgery (interview data)

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scrimin S, Haynes M, Altoe G, Bornstein MH, Axia G. Anxiety and stress in mothers and fathers in the 24 h after their child's surgery. Child Care Health Dev. 2009 Mar;35(2):227-33. doi: 10.1111/j.1365-2214.2008.00920.x. PMID 19228156
- [Background] Landier M, Villemagne T, Le Touze A, Braik K, Meignan P, Cook AR, Morel B, Lardy H, Binet A. The position of a written document in preoperative information for pediatric surgery: A randomized controlled trial on parental anxiety, knowledge, and satisfaction. J Pediatr Surg. 2018 Mar;53(3):375-380. doi: 10.1016/j.jpedsurg.2017.04.009. Epub 2017 Apr 21. PMID 28456425
- [Background] Landolt MA, Boehler U, Schwager C, Schallberger U, Nuessli R. Post-traumatic stress disorder in paediatric patients and their parents: an exploratory study. J Paediatr Child Health. 1998 Dec;34(6):539-43. doi: 10.1046/j.1440-1754.1998.00303.x. PMID 9928646
- [Background] Piira T, Sugiura T, Champion GD, Donnelly N, Cole AS. The role of parental presence in the context of children's medical procedures: a systematic review. Child Care Health Dev. 2005 Mar;31(2):233-43. doi: 10.1111/j.1365-2214.2004.00466.x. PMID 15715702
- [Background] Malik F, Marwaha R. Developmental Stages of Social Emotional Development in Children. 2022 Sep 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK534819/ PMID 30521240
- [Background] Habre W, Disma N, Virag K, Becke K, Hansen TG, Johr M, Leva B, Morton NS, Vermeulen PM, Zielinska M, Boda K, Veyckemans F; APRICOT Group of the European Society of Anaesthesiology Clinical Trial Network. Incidence of severe critical events in paediatric anaesthesia (APRICOT): a prospective multicentre observational study in 261 hospitals in Europe. Lancet Respir Med. 2017 May;5(5):412-425. doi: 10.1016/S2213-2600(17)30116-9. Epub 2017 Mar 28. PMID 28363725